CLINICAL TRIAL: NCT00676715
Title: Phase II, Multicenter, Randomized, Parallel-Group, Partially Blinded, Placebo and Avonex Controlled Dose Finding Study to Evaluate the Efficacy As Measured by Brain MRI Lesions, and Safety of 2 Dose Regimens of Ocrelizumab in Patients With RRMS
Brief Title: A Study of the Efficacy and Safety of Ocrelizumab in Patients With Relapsing-Remitting Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT4422g; 2007-006338-32 (EudraCT Number); WA21493 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — ocrelizumab; Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo (Placebo Comparator): Participants received two intravenous (IV) infusions of matching placebo separated by 14 days in Cycle 1, followed by two infusions of ocrelizumab 300 mg separated by 14 days in cycle 2. A single infusion of ocrelizumab 600 mg was administered on Day 1 of cycles 3 and 4. Each cycle was of 168 days.
  Interventions: Drug: Placebo
- Ocrelizumab 600 mg (Experimental): Participants two IV infusions of ocrelizumab 300 mg separated by 14 days in Cycle 1, followed by an infusion of ocrelizumab 600 mg on Day 1 and an infusion of placebo on Day 15 of Cycle 2. A single infusion of ocrelizumab 600 mg was administered on Day 1 of Cycles 3 and 4. Each cycle was of 168 days.
  Interventions: Drug: Ocrelizumab
- Ocrelizumab 1000 mg (Experimental): Participants received two IV infusions of ocrelizumab 1000 mg separated by 14 days in Cycle 1, followed by an infusion of ocrelizumab 1000 mg on Day 1 and an infusion of placebo on Day 15 of Cycle 2. A single infusion of ocrelizumab 1000 mg was administered on Day 1 of Cycle 3 and a single infusion of ocrelizumab 600 mg was administered on Day 1 of Cycle 4. Each cycle was of 168 days.
  Interventions: Drug: Ocrelizumab
- Avonex (Active Comparator): Participants received weekly intramuscular injections of Avonex 30 microgram (mcg) in Cycle 1, followed by two infusions of OCR 300 mg separated by 14 days in Cycle 2. A single infusion of ocrelizumab 600 mg was administered on Day 1 of Cycles 3 and 4. Each cycle was of 168 days.
  Interventions: Drug: Avonex

INTERVENTIONS:
Drug: Placebo — Placebo matching to ocrelizumab administered as IV infision in Cycle 1 Day 1.
  Arms: Placebo
Drug: Ocrelizumab — Ocrelizumab 300 mg was administered in cycle 1 followed by an infusion of ocrelizumab 600 mg on Day 1. A single infusion of ocrelizumab 600 mg was administered on Day 1 of cycles 3 and 4.
  Other Names: RO4964913
  Arms: Ocrelizumab 1000 mg; Ocrelizumab 600 mg
Drug: Avonex — Avonex was administered weekly intramuscular injections of 30 mcg in cycle 1 Day 1.
  Other Names: Interferon-beta-alpha1
  Arms: Avonex

SUMMARY:
This is a phase II, multicenter, randomized, parallel-group, partially blinded, placebo and Avonex (interferon beta-1a) controlled dose finding study to evaluate the efficacy as measured by brain MRI lesions, and safety of 2 dose regimens of ocrelizumab in participants with Relapsing Remitting Multiple Sclerosis (RRMS).

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and to be compliant with the schedule of protocol assessments
* Relapsing-remitting multiple sclerosis (MS)
* Ages 18-55 years inclusive
* For sexually active female and male participants of reproductive potential, use of reliable means of contraception

Exclusion Criteria:

* Secondary or primary progressive multiple sclerosis at screening
* Incompatibility with MRI
* Contra-indications to or intolerance of oral or IV corticosteroids
* Known presence of other neurologic disorders
* Pregnancy or lactation
* Lack of peripheral venous access
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Significant, uncontrolled disease, such as cardiovascular, pulmonary, renal, hepatic, endocrine or gastrointestinal
* Congestive heart failure
* Known active bacterial, viral, fungal, mycobacterial infection or other infection or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks prior to screening or oral antibiotics within 2 weeks prior to screening
* History or known presence of recurrent or chronic infection
* History of cancer, including solid tumors and hematological malignancies (except basal cell, in situ squamous cell carcinomas of the skin, and in situ carcinoma of the cervix of the uterus that have been excised and resolved)
* History of alcohol or drug abuse within 24 weeks prior to randomization
* History of or currently active primary or secondary immunodeficiency
* History of coagulation disorders
* Treatment with any investigational agent within 4 weeks of screening
* Receipt of a live vaccine within 6 weeks prior to randomization
* Incompatibility with Avonex use
* Previous treatment with rituximab
* Previous treatment with lymphocyte-depleting therapies except mitoxantrone
* Treatment with lymphocyte trafficking blockers within 24 weeks prior to randomization
* Treatment with beta interferons, glatiramer acetate, IV immunoglobulin, plasmapheresis, or immunosuppressive therapies within 12 weeks prior to randomization
* Systemic corticosteroid therapy within 4 weeks prior to randomization

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2008-07-17 (Actual); Primary Completion 2012-03-09 (Actual); Study Completion 2023-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (84):
- United States (26):
  - Phoenix Neurological Associates Ltd, Phoenix, Arizona
  - Barrow Neurological Institute, Phoenix, Arizona
  - East Bay Physicians Med Group;Sutter East Bay Med Foundation, Berkeley, California
  - University of California San Francisco, San Francisco, California
  - Advanced Neurology of Colorado, LLC, Fort Collins, Colorado
  - Bradenton Research Center, Bradenton, Florida
  - MS Center of Vero Beach, Vero Beach, Florida
  - Shepherd Center; Multiple Sclerosis Center, Atlanta, Georgia
  - University of Chicago; Neurology, Chicago, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - John Hopkins University, Baltimore, Maryland
  - Michigan Institute for Neurological Disorders, Farmington Hills, Michigan
  - Dartmouth-Hitchcock Medical Center; Dept of Neurology, Lebanon, New Hampshire
  - Columbia University Medical Center; The Neurological Institute of New York, New York, New York
  - Island Neurological Associates, P.C., Plainview, New York
  - Suny At Stony Brook; Department Of Neurology, Stony Brook, New York
  - The Neurological Institute PA, Charlotte, North Carolina
  - Clinical Research of Winston Salem, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Med Ctr; MS Center, Columbus, Ohio
  - Legacy Health System; Clinical Research & Tech Ctr, Tualatin, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Integra Clinical Research, Llc, San Antonio, Texas
  - Fletcher Allen Health Care/University of Vermont, Burlington, Vermont
  - University of Virginia - Fontain Research Park, Charlottesville, Virginia
- UZ Antwerpen, Edegem, Belgium
- Bulgaria (6):
  - First MHAT; Clinic of Neurology, Sofia
  - Shat of Cardiovascular Diseases; Clinic of Neurology, Sofia
  - ACIBADEM CITY CLINIC TOKUDA HOSPITAL EAD; Clinic of Neurology and Sleep Medicine, Sofia
  - UMHAT Tzaritza Yoanna Sofia; CLINIC OF NEUROLOGY, Sofia
  - CCB Medical institute, Ministry of Interior Sofia; CLINIC OF NEUROLOGY, Sofia
  - Military Medical Academy; Neurology, Sofia
- Canada (3):
  - Uni of British Columbia Hospital; Ms Clinical Research Group, Vancouver, British Columbia
  - St. Michael'S Hospital, Toronto, Ontario
  - McGill University; Montreal Neurological Institute; Neurological and Psychiatric, Montreal, Quebec
- Czechia (4):
  - Fakultni Nemocnice Ostrava; Klinika hematoonkologie FNO a LF OU, Ostrava
  - Krajska Nemocnice Pardubice Neurologicka Klinika, Pardubice
  - Fakultni nemocnice Motol; Neurologicka klinika, Prague
  - Nemocnice Teplice; Neurologicke Oddeleni - Ms Centrum, Teplice
- Aarhus Universitetshospital; Neurologisk Afd. F, Skleroseklinikken, Aarhus N, Denmark
- France (4):
  - Hopital Pellegrin-CHU de Bordeaux; Service de Neurologie, Bordeaux
  - CHU De Caen; Service De Neurologie Dejerine, Caen
  - Hopital Gabriel Montpied CHU de Clermont-Ferrand; Service de Neurologie B, Clermont-Ferrand
  - CHU De Nimes, Hopital Caremeau; Service De Neurologie Du Prof. Pierre Labauge, Nîmes
- Germany (4):
  - St. Joseph-Krankenhaus, Berlin
  - Jüdisches Krankenhaus Berlin; Abteilung fur Neurologie, Berlin
  - Asklepios Klinik Nord-Heidberg; Neurologie, Hamburg
  - Universitatsklinikum Marburg; Zentrum für Nervenheilkunde, Klinik für Psychiatrie+Psychotherapie, Marburg
- Ospedale S.Andrea-Universita di Roma; Centro Sclerosi Multipla, Rome, Lazio, Italy
- Mexico (4):
  - Hospital CIMA, Sta. Engracia, Monterrey, Nuevo León
  - Instituto Biomedico De Investigacion A.C., Aguascalientes
  - Unidad de Investigacion CIMA SC, Chihuahua City
  - Hospital Cima Chihauhau, Chihuahua City
- Romania (2):
  - Spitalul Clinic Colentina; Clinica de Neurologie, Bucharest
  - Spitalul Clinic Judetean de Urgenta Targu Mures; Clinica Neurologie, Târgu Mureş
- Russia (6):
  - Central Clinical Hospital #2 N.A. Semashko OAO RJHD, Moskva, Moscow Oblast
  - Municipal City Hospital #33; Neurology, Nizhny Novgorod, Niznij Novgorod
  - SHI Sverdlovsk Regional Clinical Hospital #1;Neurology, Yekaterinburg, Sverdlovsk Oblast
  - LLC Research Medical Complex Vashe Zdorovie, Kazan', Tatarstan Republic
  - Regional Multiple Sclerosis Centre b/o CC ECM Neftyanik; Neurology, Tyumen, Tyumen Oblast
  - MRC for Oncology and Neurology; Neurology, Novosibirsk
- Serbia (3):
  - Clinical Center of Serbia; Institute of Neurology, Belgrade
  - Clinical Center Nis; Clinic for Mental Health, Niš
  - Clinic of Neurology, Nova Sad
- Slovakia (5):
  - Fakultna Nemocnica F. D. Roosevelta; Ii. Neurologicka Klinika Szu, Banská Bystrica
  - Fakultna Nemocnica, Pracovisko Stare Mesto; Neurology, Bratislava
  - Fakultna Nemocnica Paterua, Pracovisko Trieda Snp1 Kosice; Neurologicka Klinika, Košice
  - Fakultna Nemocnica Nitra; Neurologicka Klinika, Nitra
  - Nemocnica s Poliklinikou Spisska Nova Ves, a.s., Spišská Nová Ves
- Spain (6):
  - Hospital Universitari Vall d'Hebron; Servicio de Neumo-Inmunologia, Barcelona
  - Hospital Clinic i Provincial; Servicio de Neurologia, Barcelona
  - Hospital Ramon y Cajal; Servicio de Neurologia, Madrid
  - Hospital Regional Universitario Carlos Haya; Servicio de Neurologia, Málaga
  - Hospital Universitario Virgen Macarena; Servicio de Neurologia, Seville
  - Hospital Universitario La Fe; Unidad de Esclerosis Multiple, Valencia
- Universitätsspital Basel; Neurologie, Basel, Switzerland
- Ukraine (4):
  - Ams of Ukraine; Inst. of Neurology, Psychiatry & Narcology, Kharkiv
  - City Clin.Hosp #4; Dept. of Neurology, Kyiv
  - Ukr.State Inst. of Med and Social Probl. Disab; Dept of Neur and Border states, Propetrovsk
  - Vin.Reg.Psych.Hosp.N.A Yuschenko O.I., Vnmu N.A. Pyrogov; Department of Nervous Diseases, Vinnytsia
- United Kingdom (3):
  - Walton Centre NHS Foundation Trust, Neuroscience Research Centre; CLINICAL TRIALS UNIT, Liverpool
  - Uni Hospital Queens Medical Centre; Neurology, Nottingham
  - Royal Hallamshire Hospital; Neurology, Sheffield

REFERENCES:
- [Derived] Kappos L, Li D, Calabresi PA, O'Connor P, Bar-Or A, Barkhof F, Yin M, Leppert D, Glanzman R, Tinbergen J, Hauser SL. Ocrelizumab in relapsing-remitting multiple sclerosis: a phase 2, randomised, placebo-controlled, multicentre trial. Lancet. 2011 Nov 19;378(9805):1779-87. doi: 10.1016/S0140-6736(11)61649-8. Epub 2011 Oct 31. PMID 22047971

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 220 participants were randomized, of which 218 received study treatment. Participants took part in the study at 79 investigative sites across 18 countries from July 17, 2008, to November 08, 2023.
Pre-assignment Details: The study consisted of a 96-week Treatment Period (TP) followed by a Treatment-free period (TFP). Participants who completed both TP & TFP (at least Week 120) were invited to participate in the optional Open-label Extension (OLE) period.
Groups:
- Placebo / Ocrelizumab 600 mg: In the Treatment Period, participants received placebo as, intravenous (IV) infusion on Days 1 and 15 of Cycle 1 ( 1 Cycle = 168 days ), followed by ocrelizumab, 300 milligrams (mg), IV, on Days 1 and 15 of Cycle 2. Participants then received ocrelizumab, 600 mg, IV, on Day 1 of Cycles 3 and 4. Participants who completed the TP then entered the TFP which was of variable duration. Participants who completed the TP and the TFP (at least through Week 120) and opted to enroll in the OLE period received ocrelizumab, 300 mg, IV, on Days 1 and 15 of Cycle 5 followed by a single infusion of ocrelizumab, 600 mg, every 24 weeks (Q24W).
- Ocrelizumab 600 mg / Ocrelizumab 600 mg: In the Treatment Period, participants received ocrelizumab 300 mg as IV infusion on Days 1 and 15 of Cycle 1 ( 1 Cycle = 168 days ), followed by ocrelizumab, 600 mg, IV, on Day 1 and placebo IV on Day 15 of Cycle 2. Participants then received ocrelizumab, 600 mg, IV, on Day 1 of Cycles 3 and 4. Participants who completed the TP then entered the TFP which was of variable duration. Participants who completed the TP and the TFP (at least through Week 120) and opted to enroll in the OLE period received ocrelizumab, 300 mg, IV, on Days 1 and 15 of Cycle 5 followed by a single infusion of ocrelizumab, 600 mg, Q24W.
- Ocrelizumab 1000 mg/ Ocrelizumab 600 mg: In the Treatment Period, participants received ocrelizumab 1000 mg as IV infusion on Days 1 and 15 of Cycle 1 ( 1 Cycle = 168 days ), followed by ocrelizumab, 1000 mg IV, on Day 1 and placebo IV on Day 15 of Cycle 2. Participants then received ocrelizumab, 1000 mg, IV, on Day 1 of Cycle 3 and ocrelizumab, 600 mg, IV, on Day 1 of Cycle 4. Participants who completed the TP then entered the TFP which was of variable duration. Participants who completed the TP and the TFP (at least through Week 120) and opted to enroll in the OLE period received ocrelizumab, 300 mg, IV, on Days 1 and 15 of Cycle 5 followed by a single infusion of ocrelizumab, 600 mg, Q24W.
- Avonex / Ocrelizumab 600 mg: In the Treatment Period, participants received Avonex 30 micrograms (mcg) as intramuscular (IM) injection once every week of Cycle 1 ( 1 Cycle = 168 days ), followed by ocrelizumab, 300 mg, IV, on Days 1 and 15 of Cycle 2. Participants then received ocrelizumab, 600 mg, IV, on Day 1 of Cycles 3 and 4. Participants who completed the TP then entered the TFP which was of variable duration. Participants who completed the TP and the TFP (at least through Week 120) and opted to enroll in the OLE period received ocrelizumab, 300 mg, IV, on Days 1 and 15 of Cycle 5 followed by a single infusion of ocrelizumab, 600 mg, Q24W.
Period: Treatment Period (TP)
Arm/Group | Placebo / Ocrelizumab 600 mg | Ocrelizumab 600 mg / Ocrelizumab 600 mg | Ocrelizumab 1000 mg/ Ocrelizumab 600 mg | Avonex / Ocrelizumab 600 mg
Started | 54 | 55 | 55 | 54
Completed | 48 | 46 | 43 | 46
Not Completed | 6 | 9 | 12 | 8
Not completed — Adverse Event | 0 | 3 | 2 | 2
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Failure to return | 1 | 0 | 0 | 0
Not completed — Violation of selection criteria at entry | 0 | 0 | 1 | 0
Not completed — Refused treatment/did not cooperate | 1 | 2 | 3 | 1
Not completed — Withdrew consent | 3 | 3 | 3 | 3
Not completed — Insufficient therapeutic response | 1 | 1 | 2 | 1
Not completed — Administrative | 0 | 0 | 0 | 1
Period: Treatment-free Period (TFP)
Arm/Group | Placebo / Ocrelizumab 600 mg | Ocrelizumab 600 mg / Ocrelizumab 600 mg | Ocrelizumab 1000 mg/ Ocrelizumab 600 mg | Avonex / Ocrelizumab 600 mg
Started | 49 (Participants who completed TP or withdrew from ocrelizumab entered the TFP.) | 48 (Participants who completed TP or withdrew from ocrelizumab entered the TFP.) | 50 (Participants who completed TP or withdrew from ocrelizumab entered the TFP.) | 49 (Participants who completed TP or withdrew from ocrelizumab entered the TFP.)
Completed | 35 | 32 | 30 | 35
Not Completed | 14 | 16 | 20 | 14
Not completed — Withdrawal by Subject | 3 | 3 | 4 | 5
Not completed — Reason not provided | 8 | 10 | 8 | 7
Not completed — Lost to Follow-up | 2 | 2 | 6 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Death | 1 | 1 | 1 | 0
Period: Open Label Extension (OLE)
Arm/Group | Placebo / Ocrelizumab 600 mg | Ocrelizumab 600 mg / Ocrelizumab 600 mg | Ocrelizumab 1000 mg/ Ocrelizumab 600 mg | Avonex / Ocrelizumab 600 mg
Started | 29 | 32 | 19 | 24
Completed | 22 | 21 | 11 | 14
Not Completed | 7 | 11 | 8 | 10
Not completed — Reason not provided | 3 | 4 | 1 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 4 | 3 | 3
Not completed — Adverse Event | 0 | 3 | 1 | 0
Not completed — Death | 2 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received any study drug and underwent at least one assessment of safety.
Groups:
- Placebo / Ocrelizumab 600 mg: In the Treatment Period, participants received placebo as IV infusion on Days 1 and 15 of Cycle 1 ( 1 Cycle = 168 days ), followed by ocrelizumab, 300 mg, IV, on Days 1 and 15 of Cycle 2. Participants then received ocrelizumab, 600 mg, IV, on Day 1 of Cycles 3 and 4. Participants who completed the TP then entered the TFP which was of variable duration. Participants who completed the TP and the TFP (at least through Week 120) and opted to enroll in the OLE period received ocrelizumab, 300 mg, IV, on Days 1 and 15 of Cycle 5 followed by a single infusion of ocrelizumab, 600 mg, Q24W.
- Avonex / Ocrelizumab 600 mg: In the Treatment Period, participants received Avonex 30 mcg as IM injection once every week of Cycle 1 ( 1 Cycle = 168 days ), followed by ocrelizumab, 300 mg, IV, on Days 1 and 15 of Cycle 2. Participants then received ocrelizumab, 600 mg, IV, on Day 1 of Cycles 3 and 4. Participants who completed the TP then entered the TFP which was of variable duration. Participants who completed the TP and the TFP (at least through Week 120) and opted to enroll in the OLE period received ocrelizumab, 300 mg, IV, on Days 1 and 15 of Cycle 5 followed by a single infusion of ocrelizumab, 600 mg, Q24W.
- Total: Total of all reporting groups
Arm/Group | Placebo / Ocrelizumab 600 mg | Ocrelizumab 600 mg / Ocrelizumab 600 mg | Ocrelizumab 1000 mg/ Ocrelizumab 600 mg | Avonex / Ocrelizumab 600 mg | Total
Number analyzed (Participants) | 54 | 55 | 55 | 54 | 218
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (8.8) | 35.6 (8.5) | 38.5 (8.7) | 38.1 (9.3) | 37.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 35 | 38 | 32 | 141
  Male | 18 | 20 | 17 | 22 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 7 | 7 | 26
  Not Hispanic or Latino | 48 | 49 | 48 | 47 | 192
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 2 | 1 | 6
  White | 52 | 51 | 53 | 53 | 209
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Gadolinium-Enhancing T1 Lesions Observed on Magnetic Resonance Imaging (MRI) Scans of the Brain
Description: Mean of total number of gadolinium-enhancing T1 lesions observed on MRI scans of the brain at Weeks 12, 16, 20, 24 was determined using average imputation method.
Time Frame: Week 12 to Week 24
Population: The intent-to-treat population includes all randomized participants who had received any study drug. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Placebo / Ocrelizumab 600 mg | Ocrelizumab 600 mg / Ocrelizumab 600 mg | Ocrelizumab 1000 mg/ Ocrelizumab 600 mg | Avonex / Ocrelizumab 600 mg
Number analyzed (Participants) | 54 | 51 | 52 | 52
lesions | 5.6 (12.53) | 0.6 (1.52) | 0.2 (0.65) | 6.9 (16.01)
Statistical Analysis 1: Comparison: Placebo / Ocrelizumab 600 mg vs Ocrelizumab 600 mg / Ocrelizumab 600 mg; Van Elteren test is stratified by region and presence of baseline gadolinium-enhancing lesions (absent or present); Test type: Superiority or Other; p < 0.0001, Van Elteren Test (stratified)
Statistical Analysis 2: Comparison: Placebo / Ocrelizumab 600 mg vs Ocrelizumab 1000 mg/ Ocrelizumab 600 mg; Van Elteren test is stratified by region and presence of baseline gadolinium-enhancing lesions (absent or present); Test type: Superiority or Other; p < 0.0001, Van Elteren Test (stratified)
Statistical Analysis 3: Comparison: Placebo / Ocrelizumab 600 mg vs Avonex / Ocrelizumab 600 mg; Van Elteren test is stratified by region and presence of baseline gadolinium-enhancing lesions (absent or present); Test type: Superiority or Other; p = 0.7496, Van Elteren Test (stratified)

2. Secondary Outcome: Annualized Protocol Defined Relapse Rate at Week 24
Description: Adjusted annualized relapse rate for geographical region is reported here. The relapse rate was calculated as the total number of relapses for each participant divided by the total number of patient-years.
Time Frame: Week 24
Population: The intent-to-treat population includes all randomized participants who had received any study drug.
Measure: Number (95% Confidence Interval); unit: relapses per year
Groups:
- Avonex / Ocrelizumab 600 mg: In the Treatment Period, participants received Avonex 30 mcg as IM injection every week of Cycle 1 ( 1 Cycle = 168 days ), followed by ocrelizumab, 300 mg, IV, on Days 1 and 15 of Cycle 2. Participants then received ocrelizumab, 600 mg, IV, on Day 1 of Cycles 3 and 4. Participants who completed the TP then entered the TFP which was of variable duration. Participants who completed the TP and the TFP (at least through Week 120) and opted to enroll in the OLE period received ocrelizumab, 300 mg, IV, on Days 1 and 15 of Cycle 5 followed by a single infusion of ocrelizumab, 600 mg, Q24W.
Arm/Group | Placebo / Ocrelizumab 600 mg | Ocrelizumab 600 mg / Ocrelizumab 600 mg | Ocrelizumab 1000 mg/ Ocrelizumab 600 mg | Avonex / Ocrelizumab 600 mg
Number analyzed (Participants) | 54 | 55 | 55 | 54
relapses per year | 0.557 [0.370 to 0.839] | 0.127 [0.054 to 0.299] | 0.213 [0.110 to 0.414] | 0.364 [0.220 to 0.602]
Statistical Analysis 1: Comparison: Placebo / Ocrelizumab 600 mg vs Ocrelizumab 600 mg / Ocrelizumab 600 mg; Poisson model was fitted for adjusting for geographic region only; Test type: Superiority or Other; p = 0.0019, Poisson model
Statistical Analysis 2: Comparison: Placebo / Ocrelizumab 600 mg vs Ocrelizumab 1000 mg/ Ocrelizumab 600 mg; Poisson model was fitted for adjusting for geographic region only; Test type: Superiority or Other; p = 0.0136, Poisson model
Statistical Analysis 3: Comparison: Placebo / Ocrelizumab 600 mg vs Avonex / Ocrelizumab 600 mg; Poisson model was fitted for adjusting for geographic region only; Test type: Superiority or Other; p = 0.1814, Poisson model

3. Secondary Outcome: Percentage of Participants Who Remained Relapse Free at Week 24
Description: Percentage of participants who remained relapse free at week 24 were reported. Percentages have been rounded off to the first decimal.
Time Frame: Week 24
Population: The intent-to-treat population includes all randomized participants who had received any study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo / Ocrelizumab 600 mg | Ocrelizumab 600 mg / Ocrelizumab 600 mg | Ocrelizumab 1000 mg/ Ocrelizumab 600 mg | Avonex / Ocrelizumab 600 mg
Number analyzed (Participants) | 54 | 55 | 55 | 54
percentage of participants | 75.9 [64.5 to 87.3] | 85.5 [76.1 to 94.8] | 87.3 [78.5 to 96.1] | 77.8 [66.7 to 88.9]
Statistical Analysis 1: Comparison: Placebo / Ocrelizumab 600 mg vs Ocrelizumab 600 mg / Ocrelizumab 600 mg; Test type: Superiority or Other; p = 0.1978, Cochran-Mantel-Haenszel chi-square test; Cochran-Mantel-Haenszel (CMH) chi-square test stratified by geographical region only; Relative risk (RR) = 0.60, 95% CI 2-sided [0.27 to 1.34]
Statistical Analysis 2: Comparison: Placebo / Ocrelizumab 600 mg vs Ocrelizumab 1000 mg/ Ocrelizumab 600 mg; Test type: Superiority or Other; p = 0.1310, CMH chi-square test; CMH chi-square test stratified by geographical region only; Relative risk (RR) = 0.53, 95% CI 2-sided [0.23 to 1.22]
Statistical Analysis 3: Comparison: Placebo / Ocrelizumab 600 mg vs Avonex / Ocrelizumab 600 mg; Test type: Superiority or Other; p = 0.8206, CMH chi-square tes; CMH chi-square test stratified by geographical region only; Relative risk (RR) = 0.92, 95% CI 2-sided [0.46 to 1.84]

4. Secondary Outcome: Change From Baseline in Total Volume of T2 Lesions on MRI Scans of the Brain at Week 24
Description: Change from baseline in total volume of T2 lesions on MRI scans of the brain at Week 24 was reported.
Time Frame: Baseline, Week 24
Population: The intent-to-treat population includes all randomized participants who had received any study drug. Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses at the specified timepoints.
Measure: Mean (Standard Deviation); unit: cubic millimeter (mm^3)
Arm/Group | Placebo / Ocrelizumab 600 mg | Ocrelizumab 600 mg / Ocrelizumab 600 mg | Ocrelizumab 1000 mg/ Ocrelizumab 600 mg | Avonex / Ocrelizumab 600 mg
Number analyzed (Participants) | 47 | 51 | 53 | 49
cubic millimeter (mm^3)
  Baseline | 8950.84 (9776.261) | 13972.61 (19930.158) | 13178.30 (14271.383) | 13209.11 (17206.511)
  Change at Week 24: number analyzed (Participants) | 43 | 45 | 46 | 46
  Change at Week 24 | -112.31 (1464.206) | -878.84 (2756.839) | -600.89 (2105.964) | 1040.06 (4510.140)
Statistical Analysis 1: Comparison: Placebo / Ocrelizumab 600 mg vs Ocrelizumab 600 mg / Ocrelizumab 600 mg; Test type: Superiority or Other; p = 0.1391, Van Elteren Test (stratified); Van Elteren test is stratified by region only
Statistical Analysis 2: Comparison: Placebo / Ocrelizumab 600 mg vs Ocrelizumab 1000 mg/ Ocrelizumab 600 mg; Test type: Superiority or Other; p = 0.1596, Van Elteren Test (stratified); Van Elteren test is stratified by region only
Statistical Analysis 3: Comparison: Placebo / Ocrelizumab 600 mg vs Avonex / Ocrelizumab 600 mg; Test type: Superiority or Other; p = 0.4740, Van Elteren Test (stratified); Van Elteren test is stratified by region only

5. Secondary Outcome: Total Number of New Gadolinium-Enhancing T1 Lesions Observed by MRI Scans of the Brain
Description: Total number of new gadolinium-enhancing T1 lesions observed by MRI scans of the brain were reported.
Time Frame: Weeks 4 to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Placebo / Ocrelizumab 600 mg | Ocrelizumab 600 mg / Ocrelizumab 600 mg | Ocrelizumab 1000 mg/ Ocrelizumab 600 mg | Avonex / Ocrelizumab 600 mg
Number analyzed (Participants) | 54 | 51 | 52 | 52
lesions | 5.1 (11.99) | 0.8 (1.95) | 0.8 (2.16) | 6.2 (13.79)
Statistical Analysis 1: Comparison: Placebo / Ocrelizumab 600 mg vs Ocrelizumab 600 mg / Ocrelizumab 600 mg; Test type: Superiority or Other; p < 0.0001, Van Elteren Test (stratified); Van Elteren test is stratified by region only
Statistical Analysis 2: Comparison: Placebo / Ocrelizumab 600 mg vs Ocrelizumab 1000 mg/ Ocrelizumab 600 mg; Test type: Superiority or Other; p < 0.0001, Van Elteren Test (stratified); Van Elteren test is stratified by region only
Statistical Analysis 3: Comparison: Placebo / Ocrelizumab 600 mg vs Avonex / Ocrelizumab 600 mg; Test type: Superiority or Other; p = 0.4985, Van Elteren Test (stratified); Van Elteren test is stratified by region only

6. Secondary Outcome: Total Number of Gadolinium-Enhancing T1 Lesions
Description: Total number of gadolinium-enhancing T1 lesions from Week 4 to Week 24 were reported.
Time Frame: Weeks 4 to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Placebo / Ocrelizumab 600 mg | Ocrelizumab 600 mg / Ocrelizumab 600 mg | Ocrelizumab 1000 mg/ Ocrelizumab 600 mg | Avonex / Ocrelizumab 600 mg
Number analyzed (Participants) | 54 | 51 | 52 | 52
lesions | 8.7 (17.54) | 2.5 (5.10) | 1.8 (5.26) | 10.3 (22.15)
Statistical Analysis 1: Comparison: Placebo / Ocrelizumab 600 mg vs Ocrelizumab 600 mg / Ocrelizumab 600 mg; Test type: Superiority or Other; p = 0.0004, Van Elteren Test (stratified); Van Elteren test is stratified by region only
Statistical Analysis 2: Comparison: Placebo / Ocrelizumab 600 mg vs Ocrelizumab 1000 mg/ Ocrelizumab 600 mg; Test type: Superiority or Other; p < 0.0001, Van Elteren Test (stratified); Van Elteren test is stratified by region only
Statistical Analysis 3: Comparison: Placebo / Ocrelizumab 600 mg vs Avonex / Ocrelizumab 600 mg; Test type: Superiority or Other; p = 0.2725, Van Elteren Test (stratified); Van Elteren test is stratified by region only

ADVERSE EVENTS:
Time Frame: Up to 787 Weeks
Description: The safety population included all participants who received any study drug and underwent at least one assessment of safety. As per planned analysis adverse events from both the TP and TFP were combined and reported as participants received no interventions during the TFP. As prespecified in the protocol AEs were collected as per planned arm groups irrespective of intervention or dose level and are thus reported accordingly.
Groups:
- Placebo/Ocrelizumab 600mg: In the Treatment Period, participants received placebo as IV infusion on Days 1 and 15 of Cycle 1 (1 Cycle = 168 days), followed by ocrelizumab, 300 mg, IV, on Days 1 and 15 of Cycle 2. Participants then received ocrelizumab, 600 mg, IV, on Day 1 of Cycles 3 and 4. Participants who completed the TP then entered the TFP which was of variable duration. Participants who completed the TP and the TFP (at least through Week 120) and opted to enroll in the OLE period received ocrelizumab, 300mg, IV, on Days 1 and 15 of Cycle 5 followed by a single infusion of ocrelizumab, 600mg, Q24W.
- Ocrelizumab 600mg/Ocrelizumab 600mg: In the Treatment Period, participants received ocrelizumab 300 mg as IV infusion on Days 1 and 15 of Cycle 1 (1 Cycle = 168 days), followed by ocrelizumab, 600 mg, IV, on Day 1 and placebo IV on Day 15 of Cycle 2. Participants then received ocrelizumab, 600 mg, IV, on Day 1 of Cycles 3 and 4. Participants who completed the TP then entered the TFP which was of variable duration. Participants who completed the TP and the TFP (at least through Week 120) and opted to enroll in the OLE period received ocrelizumab, 300mg, IV, on Days 1 and 15 of Cycle 5 followed by a single infusion of ocrelizumab, 600mg, Q24W
- Ocrelizumab 1000mg/Ocrelizumab 600mg: In the Treatment Period, participants received ocrelizumab 1000 mg as IV infusion on Days 1 and 15 of Cycle 1 (1 Cycle = 168 days), followed by ocrelizumab, 1000 mg IV, on Day 1 and placebo IV on Day 15 of Cycle 2. Participants then received ocrelizumab, 1000 mg, IV, on Day 1 of Cycles 3 and 4. Participants who completed the TP then entered the TFP which was of variable duration. Participants who completed the TP and the TFP (at least through Week 120) and opted to enroll in the OLE period received ocrelizumab, 300mg, IV, on Days 1 and 15 of Cycle 5 followed by a single infusion of ocrelizumab, 600mg, Q24W.
- Avonex/Ocrelizumab 600 mg: In the Treatment Period, participants received Avonex 30 mcg as IM injection once every week of Cycle 1 (1 Cycle = 168 days), followed by ocrelizumab, 300 mg, IV, on Days 1 and 15 of Cycle 2. Participants then received ocrelizumab, 600 mg, IV, on Day 1 of Cycles 3 and 4. Participants who completed the TP then entered the TFP which was of variable duration. Participants who completed the TP and the TFP (at least through Week 120) and opted to enroll in the OLE period received ocrelizumab, 300mg, IV, on Days 1 and 15 of Cycle 5 followed by a single infusion of ocrelizumab, 600mg, Q24W.
- Ocrelizumab 600 mg Open Label Extension (OLE): Participants who opted to enroll in the OLE received two IV infusions of ocrelizumab, 300mg on Days 1 and 15 of Cycle 5, followed by a single infusion of ocrelizumab, 600mg, once Q24W
Arm/Group | Placebo/Ocrelizumab 600mg | Ocrelizumab 600mg/Ocrelizumab 600mg | Ocrelizumab 1000mg/Ocrelizumab 600mg | Avonex/Ocrelizumab 600 mg | Ocrelizumab 600 mg Open Label Extension (OLE)
All-Cause Mortality (participants affected / at risk) | 3/54 | 1/55 | 3/55 | 2/54 | 6/103
Serious Adverse Events (participants affected / at risk) | 11/54 | 17/55 | 16/55 | 16/54 | 28/103
Other Adverse Events (participants affected / at risk) | 52/54 | 47/55 | 45/55 | 45/54 | 85/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Ocrelizumab 600mg (N=54) | Ocrelizumab 600mg/Ocrelizumab 600mg (N=55) | Ocrelizumab 1000mg/Ocrelizumab 600mg (N=55) | Avonex/Ocrelizumab 600 mg (N=54) | Ocrelizumab 600 mg Open Label Extension (OLE) (N=103)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
IMMUNE THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ADRENAL CYST (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
RETINAL ARTERY OCCLUSION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INGUINAL HERNIA STRANGULATED (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SALIVARY DUCT INFLAMMATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUBILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEATH (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DRUG WITHDRAWAL SYNDROME (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
COMPLICATED APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
COVID-19 PNEUMONIA (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 6 (6)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ENCEPHALITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GINGIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEPATITIS A (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ORAL HERPES (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
TRACHEOBRONCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 3 (5)
UROSEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
AMYLASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
BLOOD POTASSIUM INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
SMEAR CERVIX ABNORMAL (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EPILEPSY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MULTIPLE SCLEROSIS PSEUDO RELAPSE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (3)
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
MUSCLE SPASTICITY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE PSYCHOSIS (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUSPECTED SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URETEROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OVARIAN MASS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UTERINE PROLAPSE (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Ocrelizumab 600mg (N=54) | Ocrelizumab 600mg/Ocrelizumab 600mg (N=55) | Ocrelizumab 1000mg/Ocrelizumab 600mg (N=55) | Avonex/Ocrelizumab 600 mg (N=54) | Ocrelizumab 600 mg Open Label Extension (OLE) (N=103)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
PALPITATIONS (Cardiac disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 3 (3)
VISION BLURRED (Eye disorders) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 3 (3)
CONSTIPATION (Gastrointestinal disorders) | 3 (3) | 3 (3) | 4 (4) | 2 (2) | 4 (4)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 4 (6) | 5 (6) | 2 (2) | 5 (7)
HAEMORRHOIDS (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (2) | 0 (0) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 2 (3) | 7 (10) | 4 (5) | 5 (5)
ASTHENIA (General disorders) | 3 (5) | 2 (2) | 2 (3) | 1 (1) | 3 (3)
CHILLS (General disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
FATIGUE (General disorders) | 5 (8) | 7 (7) | 11 (14) | 4 (4) | 8 (12)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 2 (2) | 2 (2) | 11 (15) | 3 (3)
OEDEMA PERIPHERAL (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
PYREXIA (General disorders) | 3 (3) | 8 (8) | 3 (4) | 2 (2) | 11 (12)
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 4 (4)
SEASONAL ALLERGY (Immune system disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
BRONCHITIS (Infections and infestations) | 7 (12) | 4 (4) | 6 (11) | 2 (2) | 10 (17)
COVID-19 (Infections and infestations) | 12 (13) | 7 (8) | 5 (5) | 2 (4) | 26 (30)
CYSTITIS (Infections and infestations) | 4 (5) | 2 (4) | 5 (6) | 0 (0) | 4 (4)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 5 (5)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 5 (7) | 1 (1) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
INFLUENZA (Infections and infestations) | 7 (8) | 4 (4) | 7 (11) | 4 (5) | 10 (14)
NASOPHARYNGITIS (Infections and infestations) | 10 (15) | 15 (32) | 12 (25) | 9 (25) | 20 (41)
ORAL HERPES (Infections and infestations) | 4 (17) | 3 (7) | 2 (3) | 4 (5) | 6 (18)
PHARYNGITIS (Infections and infestations) | 6 (7) | 3 (6) | 1 (1) | 3 (4) | 5 (6)
PNEUMONIA (Infections and infestations) | 3 (5) | 1 (1) | 3 (4) | 1 (1) | 7 (10)
PYELONEPHRITIS (Infections and infestations) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (18) | 5 (8) | 2 (5) | 3 (5) | 8 (9)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 2 (2) | 3 (6) | 1 (1) | 1 (1) | 3 (4)
SINUSITIS (Infections and infestations) | 5 (7) | 4 (4) | 3 (4) | 2 (2) | 5 (6)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 (17) | 14 (25) | 11 (26) | 7 (10) | 15 (32)
URINARY TRACT INFECTION (Infections and infestations) | 14 (29) | 10 (24) | 15 (39) | 10 (17) | 23 (58)
VAGINAL INFECTION (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
VIRAL INFECTION (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
CONTUSION (Injury, poisoning and procedural complications) | 2 (3) | 3 (3) | 3 (3) | 1 (1) | 3 (3)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 29 (63) | 25 (60) | 29 (60) | 20 (33) | 23 (39)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 5 (6) | 1 (1) | 1 (1)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
THERMAL BURN (Injury, poisoning and procedural complications) | 3 (4) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 5 (5)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 (15) | 9 (10) | 5 (8) | 5 (8) | 13 (18)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 9 (11) | 5 (7) | 4 (5) | 7 (9) | 6 (7)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 3 (4) | 1 (1) | 4 (4)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 3 (3)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 7 (11) | 2 (2) | 8 (10) | 2 (2) | 8 (10)
DIZZINESS (Nervous system disorders) | 5 (6) | 4 (4) | 4 (6) | 1 (1) | 2 (2)
HEADACHE (Nervous system disorders) | 15 (33) | 9 (16) | 10 (14) | 12 (19) | 7 (11)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 2 (3) | 5 (5) | 3 (4) | 3 (3)
MIGRAINE (Nervous system disorders) | 5 (6) | 4 (6) | 2 (2) | 1 (1) | 4 (5)
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 26 (70) | 19 (39) | 21 (72) | 29 (58) | 28 (68)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 4 (4) | 5 (5) | 1 (1) | 0 (0)
SCIATICA (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
SYNCOPE (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 3 (3) | 5 (7) | 3 (3) | 6 (6) | 4 (4)
DEPRESSION (Psychiatric disorders) | 2 (2) | 7 (8) | 5 (5) | 4 (5) | 5 (5)
INSOMNIA (Psychiatric disorders) | 2 (3) | 3 (4) | 9 (12) | 1 (1) | 4 (4)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 4 (5)
RENAL CYST (Renal and urinary disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (5) | 3 (3) | 4 (4) | 5 (7)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 3 (3) | 1 (1) | 2 (3)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 3 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 2 (2) | 1 (2) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3) | 4 (4) | 4 (4) | 3 (3)
SKIN LESION (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
HYPERTENSION (Vascular disorders) | 4 (4) | 6 (7) | 0 (0) | 1 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsorâ€™s intellectual property rights.